CLINICAL TRIAL: NCT06098612
Title: PET Imaging Evaluation of [11C]SY08
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Changning Wang, Associate Professor, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023P002302
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Parkinson's Disease; Multiple System Atrophy; Dementia With Lewy Bodies; Healthy Controls
MeSH Terms: conditions — Parkinson Disease; Multiple System Atrophy; Lewy Body Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- evaluation of alpha synuclein aggregates in the brain (Experimental)
  Interventions: Drug: C11-SY08

INTERVENTIONS:
Drug: C11-SY08 — a PET imaging agent

SUMMARY:
The overall goal of the proposed research is to evaluate the use of [11C]SY08 as a PET radiotracer for aggregated alpha synuclein (αS) in individuals with Parkinson's disease (PD), Multiple system atrophy (MSA), Dementia with Lewy Bodies (DLB) and healthy controls.

The purpose of this study is to evaluate the use of [11C]SY08 as a PET radiotracer for αS fibrils in individuals with PD, MSA, DLB and healthy controls. The specific aims of the current study are:

1. To determine brain uptake, distribution, and kinetics of [11C]SY08 in healthy individuals.
2. To determine brain uptake, distribution, and kinetics of [11C]SY08 in patients with alpha synuclein aggregates in the brain, including PD, DLB and MSA.
3. To determine human dosimetry of [11C]SY08 in healthy individuals

An intravenous bolus injection of [11C]SY08 will be administered per subject for brain PET imaging.

ELIGIBILITY:
Inclusion Criteria:

* General Inclusion criteria, all subjects must:

  1. Age 50-80
  2. Be able to provide written informed consent or assent
  3. Be able to read, speak and understand English (The investigators do not have the resources necessary to properly study non-English speaking patients in this study, given that translation and validation of the assessment tools would be necessary)
  4. Be willing and able to participate in one PET/MRI scanning session

Additional Inclusion criteria for PD patients, subjects must:

1. Have an existing diagnosis of idiopathic PD, using consensus criteria
2. Stable medications for at least 30 days
3. Hoehn and Yahr stage I-IV
4. A study partner who can answer questions pertaining to daily functioning

Additional Inclusion criteria for MSA patients, subjects must:

1. Have an existing diagnosis of MSA, using consensus criteria
2. Stable medications for at least 30 days
3. MSAp or MSAc
4. A study partner who can answer questions pertaining to daily functioning

Additional Inclusion criteria for DLB patients, subjects must:

1. Have an existing diagnosis of probable DLB, using consensus criteria
2. Stable medications for at least 30 days
3. Clinical Dementia Rating Scale (CDR) < 0.5
4. A study partner who can answer questions pertaining to daily functioning

Exclusion Criteria:

* General Exclusion Criteria (All Subjects)

  1. History of vascular risk factors (e.g. hypertension, hyperlipidemia), if not well-controlled
  2. Major psychiatric disease (e.g.schizophrenia)
  3. History of stroke
  4. Focal brain lesions on MRI scans
  5. History of other major illnesses including, but not limited to, major kidney or liver problems or significant neurological illness
  6. Recent surgery that is deemed major by our reviewing physician or nurse practitioner within the past 6 months
  7. History of head trauma (as defined as having any insults to the brain that may have resulted from an external mechanical force, such as rapid acceleration or deceleration, impact, blast waves, or penetration by a projectile)
  8. Impaired elimination (as defined as having problems with urination) unless being managed
  9. Past or present diagnosis of bipolar disorder or other Axis I diagnosis, (treated depression is allowed)
  10. Any present substance abuse including drug/alcohol abuse
  11. Inability to lie flat on camera bed for up to 90 min
  12. Pregnancy or breastfeeding
  13. Metallic foreign bodies that would be affected by the MRI magnet, or fear of enclosed spaces likely to make the subject unable to undergo an MRI scan
  14. Recent exposure to radiation (i.e., PET from other research) that, when combined with this study, would be above the allowable limits (50 milliSieverts)

General MR and PET safety exclusion criteria listed below

1. Ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, metallic tattoos anywhere on the body, tattoos near the eye, steel implants, ferromagnetic objects such as jewelry or metal clips in clothing
2. Electrical implants such as cardiac pacemakers or perfusion pumps
3. Pre-existing medical conditions including a likelihood of developing seizures or claustrophobic reactions, and any greater than normal potential for cardiac arrest
4. Is unable to lie comfortably on a bed inside a PET camera with their head in the field of view for 60 to 90 minutes as assessed by physical examination and medical history (e.g. back pain, arthritis)
5. Pregnancy: A negative serum pregnancy test is required on the day of the PET procedure in women of child bearing potential
6. Body weight of > 300 lbs (weight limit of the MRI table)
7. Breast feeding mothers

Exclusion Criteria for Subjects Undergoing Blood Draws Through an Arterial Line During PET Scan

1. An abnormal result on the modified Allen's test on both hands
2. Raynaud syndrome
3. Bleeding disorder
4. Use of anticoagulants such as Coumadin, Plavix or Lovenox
5. An allergy to Lidocaine

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
brain uptake evaluation | up tp 120 minutes
  The investigators will use SUV or SUV to evaluate brain uptake

CONTACTS AND LOCATIONS:
Locations (1):
- MGH, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No